CLINICAL TRIAL: NCT05183529
Title: Monitoring Vital Signs With a Wireless Ingestible Device in Subjects Undergoing Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celero Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-002
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Sleep
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing polysomnography (Experimental)
  Interventions: Device: Vitals Monitoring Pill System

INTERVENTIONS:
Device: Vitals Monitoring Pill System — The Celero Vitals Monitoring Pill (VM Pill) uses 3 axis accelerometry to measure physiological signals from within the GI tract.

SUMMARY:
This Minimal Risk study is designed to evaluate the ability of the Celero ingestible Vitals Monitoring Pill (i.e., VM Pill) to measure respiration from within the gastrointestinal tract, in addition to performing an exploratory comparative analysis of data collected by the VM Pill and data collected from clinical monitoring sensors as part of polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals ages 18 - 65 inclusive who are indicated for a polysomnography study.

Exclusion Criteria:

* Patients with a history of abdominal surgery and/or any condition that may impact the GI tract, including but not limited to:

  * Constipation
  * Esophageal stricture
  * Esophagitis
  * Gastritis
  * Gastric ulcers
  * Peptic ulcer
  * Gallstones
  * Celiac Disease
  * Crohn's Disease
  * Ulcerative Colitis
  * Irritable Bowel Syndrome
  * Diverticulitis
  * Colorectal cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the ability of the VM Pill to monitor respiration from within the GI tract | During polysomnography
  Mean absolute error between respiratory rate measured by the VM Pill and respiratory rate measured by PSG monitoring equipment during periods of normal breathing while the patient is sleeping or at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Kupec, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States